CLINICAL TRIAL: NCT00305344
Title: Transfusion of Autologous Umbilical Cord Blood to Reverse Hyperglycemia in Children With Type 1 Diabetes - A Pilot Study
Brief Title: Umbilical Cord Blood Infusion to Treat Type 1 Diabetes
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1-2005-362; GCRC 593 (Other: General Clinical Research Center); UF IRB-01 125-2004 (Other: UF Institutional Review Board)
Record Dates: First submitted 2006-03-17; First posted 2006-03-21 (Estimated); Results first posted 2012-07-10 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus; Umbilical Cord; Regeneration; Insulin; Islets of Langerhans
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Cord Blood (Active Comparator): Umbilical Cord Blood
  Interventions: Procedure: Autologous Umbilical Cord Blood Transfusion; Biological: Cord blood

INTERVENTIONS:
Procedure: Autologous Umbilical Cord Blood Transfusion — Cord Blood infusion
  Other Names: Cord Blood
Biological: Cord blood — Develop Cord blood vaccine
  Other Names: Vaccine

SUMMARY:
While this study is now completely enrolled, we do hope to develop a "next generation" cord blood based study sometime in early 2009. Please continue to contact us if you have a child with newly diagnosed Type 1 Diabetes (T1D) who alo has their OWN cord blood in storage.

DETAILED DESCRIPTION:
Objective:

Our goal is to transfuse autologous umbilical cord blood into 23 children with T1D in an attempt to re-establish immune tolerance and perhaps regenerate pancreatic islet insulin-producing beta cells and improve blood glucose control. As secondary goals, we aim to study the potential changes in metabolism/immune function leading to islet regeneration.

Background/Rationale:

Stem cells provide an exciting approach towards curing T1D. Autologous bone marrow transplants have been used successfully for patients undergoing high dose chemotherapy, and for a variety of cancers and autoimmune disorders such as multiple sclerosis, lupus, and rheumatic disorders. Recent studies in immunodeficient mice with chemically-induced pancreatic damage have shown that bone marrow-derived stem cells preferentially home to the pancreas and may have the capacity to initiate pancreatic regeneration, thereby restoring the endothelial interactions in the pancreas and correcting the associated elevated blood sugar levels Human umbilical cord blood cells transfused into a model of amyotrophic lateral sclerosis (ALS) resulted in delayed disease progression of two to three weeks and increased lifespan. Umbilical cord blood has shown promise as an excellent source for deriving stem cell populations, and has been used successfully in transplantation for a variety of diseases, including acute lymphocytic and myeloid leukemia, lymphoma, Fanconi anemia, and sickle cell disease. Furthermore, umbilical cord blood-derived stem cells have the capacity to differentiate into a variety of non-blood cell types, including hepatocytes, neural cells, and endothelial cells. In addition, umbilical cord blood contains a greater proportion of hematopoietic stem cells than bone marrow.

In addition, cord blood contains a large number of immune cells called regulatory T cells, These regulatory T cells may be helpful in diminishing autoimmunity. The need to re-establish tolerance in patients with established autoimmunity provides another potential mechanism for cord blood as a therapy for type 1 diabetes.

Description of Project:

23 children > 1 year of age with T1D and stored umbilical cord blood are being be recruited. The cord blood will be infused into the children in the GCRC in an attempt to regenerate pancreatic islet insulin-producing beta cells and improve blood glucose control. As secondary goals, we aim to track the migration of transfused cord blood stem and study the potential changes in metabolism/immune function leading to islet regeneration.

Anticipated Outcome:

It is hoped that there will be preservation of beta cell function assessed by mixed meal stimulated C-peptide secretion. Changes in immunological markers/function may be observed

Relevance to Type I Diabetes:

Type 1 diabetes is still associated with tremendous morbidity and premature mortality. Patients require multiple daily insulin injections throughout their lives as well as close monitoring of their diet and blood sugar levels to prevent complications. Unfortunately, there is presently no permanent cure for diabetes. Whole pancreas or islet cell transplantation is available only to a very limited number of patients and necessitates potential lifelong immunosuppressive therapy. The need to find a cure for T1D cannot be overstated -autologous stem cell transfusions either with their potential to differentiate into islet cells or provide immune tolerance that leads to islet regeneration appear to be a safe and potentially viable option.

ELIGIBILITY:
Inclusion Criteria:

1. Must have a diagnosis of T1D and have stored umbilical cord blood in an AABB and/or FACT accredited cord bank.
2. TID diagnosis will be defined as having a clear history of polydipsia, polyphagia, polyuria, and weight loss consistent with a clinical diagnosis, diagnosis will mot be based solely upon the presence of autoantibodies.
3. Cord blood meets all selection and testing criteria (see below).
4. Able to complete mixed meal tolerance / glucagon stimulation test.
5. Normal screening values for CBC, Renal function and electrolytes (BMP).
6. Willing to comply with intensive diabetes management

Exclusion Criteria:

1. Complicating medical issues that would interfere with blood drawing or monitoring.
2. Chronic use of steroids or other immunosuppressive agents for other conditions.
3. Positive infectious disease markers from mothers' blood or cord at time of collection (See below for details).
4. Any evidence of illness on planned infusion date (i.e. fever >38.5 C, vomiting, diarrhea, wheezing, or crackles).

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2005-04; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Haller, MD, Principal Investigator — University of Florida; Desmond A Schatz, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Result] Haller MJ, Wasserfall CH, Hulme MA, Cintron M, Brusko TM, McGrail KM, Sumrall TM, Wingard JR, Theriaque DW, Shuster JJ, Atkinson MA, Schatz DA. Autologous umbilical cord blood transfusion in young children with type 1 diabetes fails to preserve C-peptide. Diabetes Care. 2011 Dec;34(12):2567-9. doi: 10.2337/dc11-1406. Epub 2011 Oct 19. PMID 22011412
- [Result] Haller MJ, Wasserfall CH, McGrail KM, Cintron M, Brusko TM, Wingard JR, Kelly SS, Shuster JJ, Atkinson MA, Schatz DA. Autologous umbilical cord blood transfusion in very young children with type 1 diabetes. Diabetes Care. 2009 Nov;32(11):2041-6. doi: 10.2337/dc09-0967. PMID 19875605

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 23 total subjects were enrolled.
Pre-assignment Details: Patients with autologous cord blood in private storage facilities were eligible. No eligible patients were excluded.
Groups:
- Cord Blood Recipient: Umbilical Cord Recipient
Period: Overall Study
Arm/Group | Cord Blood Recipient
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cord Blood Recipient
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 5.1 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Children With T1D Underwent a Single Autologous UCB Transfusion
Description: All participants were monitored for 2 years. Baseline and post-infusion mixed meal tolerance tests were performed to determine whether autologous cord blood infusion preserved endogenous insulin production. The change in median area under the curve for C-peptide (measure of insulin production) from baseline to to 2 years during a 2 hour mixed meal tolerance test was used as the primary outcome measure and was reported in ng/ml/120 minutes
Time Frame: Baseline to Year 2
Population: All participants received their own autologous umbilical cord blood (UCB)
Measure: Median (Inter-Quartile Range); unit: ng /ml /120 min
Groups:
- Recipients Receiving Cord Blood: Children with type 1 diabetes who underwent an autologous cord blood infusion
Arm/Group | Recipients Receiving Cord Blood
Number analyzed (Participants) | 23
ng /ml /120 min | -0.6 [-1.0 to -0.37]
Statistical Analysis 1: Comparison: Recipients Receiving Cord Blood; Null hypothesis: there will be no difference between AUC C-peptide at baseline and 1 or 2 years post cord blood infusion; Test type: Superiority or Other; p > 0.05, Fisher Exact

ADVERSE EVENTS:
Time Frame: 2 years
Groups:
- Cord Blood Recipients: Children with type 1 diabetes who underwent an autologous cord blood infusion
Arm/Group | Cord Blood Recipients
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

LIMITATIONS AND CAVEATS:
Small sample size. No randomized control group

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No